CLINICAL TRIAL: NCT04263727
Title: A Longitudinal Observational Study of Patients With Chronic Disease
Brief Title: A Study of Patients With Chronic Disease
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision to terminate study
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-RWE
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-11

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Idiopathic Pulmonary Fibrosis; IPF; COPD; Respiratory Disease
Keywords: IPF; COPD; Respiratory Disease; Asthma
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Patients enrolled in TARGET-RWE may be invited to participate in the Biorepository Bank (BSB). Blood samples for biomarker and DNA assays will be collected on a voluntary basis and participation in this project will not affect participation in the main study. These samples will be shipped to a central repository for storage to use in future studies. Samples stored at the biorepository will be identified only with the participant's unique study ID number and the date the sample was obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asthma: Non-Interventional. Patients with asthma will be screened and enrolled into the active Asthma disease-specific cohort.
- Chronic Obstructive Pulmonary Disease (COPD): Non-Interventional. Patients with COPD will be screened into the inactive COPD disease-specific cohort.
- Idiopathic Pulmonary Fibrosis (IPF): Non-Interventional. Patients with IPF will be screened into the inactive IPF disease-specific cohort.

SUMMARY:
TARGET-RWE is a 10-year, international, longitudinal, observational study of patients with chronic disease designed to specifically address important clinical questions that remain incompletely answered from registration trials. The protocol will follow a master protocol design in which a shared study infrastructure supports progressive development of the registry across the spectrum of chronic diseases.

DETAILED DESCRIPTION:
The TARGET-RWE master protocol design allows shared study parameters and operational components to be organized within a centralized platform. Utilizing this platform, therapeutic area-aligned Communities with associated Disease-Specific Cohorts (DSC) can be added according to scientific merit and need to address specific research questions in patients diagnosed with chronic diseases. This design capitalizes on a shared, sustainable infrastructure across a diverse patient population, which allows for more efficient coordination and conduct than can be achieved in traditional stand-alone, independently-conducted research studies with narrowly-focused target patient populations. This master protocol design will ultimately support a dynamic program that adapts to the changing landscape of chronic disease management and allows for rapid enrollment and collection of retrospective and long-term prospective data from participants in specific disease areas of interest.

TARGET-RWE currently includes the TARGET-RWE.LUNG Community, with open DSCs for Asthma, COPD and Idiopathic Pulmonary Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children being managed or treated for a chronic disease under study. Diagnosis is based on the clinical judgement of the care provider.
* Patient is anticipated to have continued management of their chronic disease at the participating site.

Exclusion Criteria:

* Inability to provide informed assent/consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with chronic disease in the United States and Europe.
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Natural history of chronic disease under study: Characteristics of chronic diseases under study. | Up to 10 years
Natural history of chronic disease under study: Participant demographics | Up to 10 years
Natural history of chronic disease under study: Treatment use | Up to 10 years
Natural history of chronic disease under study: Disease progression | Up to 10 years
Adverse event frequency and severity | Up to 10 years

SECONDARY OUTCOMES:
Natural history of chronic disease under study: Treatment response | Up to 10 years
Time point of clinical response | Every 12 months for 10 years
Reasons for treatment discontinuation | Up to 10 years
Self-reported patient health measures: Asthma Control Test | Every 12 months for 10 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - St. Francis Medical Institute, Clearwater, Florida
  - Family Allergy & Asthma Research Institution, Louisville, Kentucky
  - University of Michigan Allergy Specialty Clinic & Food Allergy, Ann Arbor, Michigan
  - Coastal Carolina Healthcare, P.A., New Bern, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided